CLINICAL TRIAL: NCT01325402
Title: Open-Label Positron Emission Tomography Study With Selective Beta Amyloid Radioligand (18Fluor)AZD4694 to Assess the Effects of Varying Mass of AZD4694 on Radioligand Binding Parameters in Healthy Volunteers and Patients With Alzheimer's Disease
Brief Title: An Open Positron Emission Tomography Study to Assess the Effects of Varying Mass of AZD4694 on Radioligand Binding Parameters in Healthy Volunteers and Patients With Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D2750C00002; EudraCT # 2011-000095-34
Record Dates: First submitted 2011-03-21; First posted 2011-03-29 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-12

CONDITIONS: Maximum Diagnostic Mass of [18Fluor]AZD4694
Keywords: Radioligand; Alzheimers disease; Maximum Diagnostic Mass; Beta amyloid
MeSH Terms: conditions — Alzheimer Disease; Plaque, Amyloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1 Cohort 1 (Experimental): Patients with mild to moderate Alzheimer's Disease
  Interventions: Other: [18Fluor]AZD4694
- Part 1 Cohort 2 (Experimental): Patients with mild to moderate Alzheimer's Disease. To run if Maximum Detective Mass is detected in cohort 1.
  Interventions: Other: [18Fluor]AZD4694
- Part 2 (Experimental): Healthy Volunteers
  Interventions: Other: [18Fluor]AZD4694

INTERVENTIONS:
Other: [18Fluor]AZD4694 — Low mass dose below 5ug. High mass dose around 40 and 50 ug.
  Arms: Part 1 Cohort 1
Other: [18Fluor]AZD4694 — Low mass dose below 5ug. High mass dose around 20 ug.
  Arms: Part 1 Cohort 2
Other: [18Fluor]AZD4694 — Low mass dose below 5ug. High mass dose will be the Maximum Detective Mass established in the previous panels.
  Arms: Part 2

SUMMARY:
In this study different mass of the radioligand AZD4694 will be given to patients with Alzheimer's Disease and healthy volunteers to evaluate wich Mass of AZD4694 that gives the best opportunities for following disease progress and treatment effects.

DETAILED DESCRIPTION:
Open-Label Positron Emission Tomography Study with Selective Beta Amyloid Radioligand (18Fluor)AZD4694 to Assess the Effects of Varying Mass of AZD4694 on Radioligand Binding Parameters in Healthy Volunteers and Patients with Alzheimer's Disease

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index between 18 and 30 kg/m2 and weigh at least 50kg and no more than 100 kg.
* Mini Mental State Examination score >28 (healthy volunteers only)
* Mini Mental State Examination score 16-28 (Alzheimer's Disease patients only)
* Hachinski Ischemic Score =4 (Alzheimer's Disease patients only)
* Clinical diagnosis of probable Alzheimer's Disease according to National Institute of Neurology and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association criteria (Alzheimer's Disease patients only)

Exclusion Criteria:

* Significant Neurological disease or dementia, as defined clinically or by imaging, other than Alzheimer's Disease that may affect cognition or ability to complete the study (Alzheimer's Disease patients only).
* Possible, probable or definite vascular dementia in accordance with the National Institute of neurology and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders association criteria (Alzheimer's Disease patients only).
* Current major depressive disorder or other major psychiatric disorders according to Diagnostic and Statistical Manual of Mental Disorders, edition 4, American Psychiatric Association 1994 criteria (Alzheimer's disease patients only).
* Depression: Cornell Depression Rating >9 (Alzheimer's disease patients only).
* Abnormal vital signs defined as any of the following: Systolic blood pressure >180 mmHg, Diastolic blood pressure >90 mmHg, heart rate <40 or>85 beats per minute (Alzheimer's disease patients only).
* Myocardial infarction or acute coronary syndrome within the last year (Alzheimer's disease patients only).
* Had Positron Emission Tomography measurements for scientific purposes within the last 12 months.
* History of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study (healthy volunteers only).
* History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs (healthy volunteers only).
* History of previous (within the last 5 years) or ongoing psychiatric disease/condition including psychosis, affective disorder, anxiety disorder, borderline state and personality disorder according to the criteria in to Diagnostic and Statistical Manual of Mental Disorders, edition 4, American Psychiatric Association 1994, as assessed by the Mini international neuropsychiatric interview (healthy volunteers only).
* Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of Investigational Product (healthy volunteers only).
* Any clinically significant abnormalities in clinical chemistry, haematology or urinalysis results as judged by the investigator (healthy volunteers only).
* Healthy volunteers<65 years: abnormal vital signs defined as any of the following: Systolic blood pressure >140 mmHg, Diastolic blood pressure >90 mmHg, heart rate <40 or>85 beats per minute.
* Healthy volunteers≥65 years: abnormal vital signs defined as any of the following: Systolic blood pressure >160 mmHg, Diastolic blood pressure >90 mmHg, heart rate <40 or >85 beats per minute.
* Central Nervous system infarct, infection of focal lesions of clinical significance on MRI scans as judged by the investigator.

Ages: 50 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
The Maximum Diagnostic Mass by assessing the visual read out of amyloid status according to and quantification of an [18F]AZD4694 PET image in a high mass experiment compared to the image in a low mass experiment in the same subject. | Visit 3
  Measuring the maximum chemical mass not causing any significant alteration of the amyloid status (unit = micrograms)
The Maximum Diagnostic Mass by assessing the visual read out of amyloid status according to and quantification of an [18F]AZD4694 PET image in a high mass experiment compared to the image in a low mass experiment in the same subject. | Visit 4
  Measuring the maximum chemical mass not causing any significant alteration of the amyloid status (unit = micrograms)

SECONDARY OUTCOMES:
Number of Adverse Events as a measure of Safety and tolerability of [18F]AZD4694 | Range of Visits 3-5
Correlation between early uptake of [18F]AZD4694 images and cerebral blood flow images as measured by Arterial Spin Labeling Magnetic resonance imaging | Range of Screening Visit to Visit 4
Correlation between estimates of β-amyloid load in brain obtained using [18F]AZD4694 Position Emission Tomography imaging and concentrations of β-amyloid in Cerebrospinal fluid | Range of Screening Visit to Visit 4

CONTACTS AND LOCATIONS:
Overall Officials: Bjorn Paulsson, Study Director — AstraZeneca; Niels Andreasen, MD, Principal Investigator — Geriatric clinic Karolinska University Hospital Huddinge; Elisabeth Eden, MD, Principal Investigator — Quintiles Aktiebolag
Locations (2):
- Sweden (2):
  - Research Site, Stockholm
  - Research Site, Uppsala